CLINICAL TRIAL: NCT02223156
Title: Effects of Mediyoga in Patients With Paroxysmal Atrial Fibrillation-MYPAF, a Randomized Controlled Three Arms Study
Brief Title: Effects of Mediyoga in Patients With Paroxysmal Atrial Fibrillation-MYPAF
Acronym: MYPAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other); Sophiahemmet University (Other)
Responsible Party: Principal Investigator, Maria Nilsson, RN, Danderyd Hospital
Other Study IDs: DNR 2013/953-31/4
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — BNP and CRP
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- MediYoga
- Music relaxation
- No treatment

SUMMARY:
The main purpose of this study is to investigate effect of Medi Yoga on quality of life, biomedical factors and health care consumption, and to study gender differences between individuals diagnosed with paroxysmal atrial fibrillation (PAF). Furthermore, an additional purpose is to describe people's experiences of Medi Yoga and identify how Medi Yoga affects their condition.

Hypothesis Individuals with PAF exercising Medi Yoga improve their quality of life and blood pressure, heart rate and heart rate variability. Biological markers such as NT-proBNP and CRP are positively affected, and that individuals seek less medical care.

DETAILED DESCRIPTION:
Methods / materials The chosen study design is a randomized Three arms controlled trial. The study will be conducted at the Cardiology Clinic at Danderyd Hospital in Stockholm. One hundred and thirty two individuals will be included and randomized to the intervention group (yoga), Music relaxation group or control group (usual follow-up). Inclusion criteria are the diagnosis of PAF and experience of symptomatic atrial fibrillation verified by ECG in the last six months. Exclusion criteria are language difficulties, multi-diagnosis and/or cognitive dysfunction (eg, diagnoses of mental illness, dementia) who are judged not to be able to perform yoga. Individuals with persistent or permanent atrial fibrillation are also excluded.

The subjects in the intervention group will practice yoga in groups for one hour once a week for 12 weeks in the hospital, with the guidance of a trained yoga instructor. They will receive written instructions on yoga exercises and a CD record to perform the yoga program at home. Added to that, the standard treatment i.e. drugs, cardioversion or ablation. The music relaxation group will listen to Music in half an hour in a group at the hospital.The control group receives usual care.

Participants are followed for three months and the evaluation is done at baseline and after three months. During these visits quality of life will be measured with two surveys, as well as variables such as blood pressure, heart rate, biological markers (CRP , BNP) , and ECG and 24-hour ECG . Primary endpoint: quality of life. In order to obtain a five -point difference in the quality of life, 132 subjects are required to achieve a power of 80 percent (p-value 0.05), including a loss rate of 20 percent. The calculation is based on the results of Substudy I. Analytical methods that will be used are: multivariate analyzes eg logistic regression, MANOVA, etc. and univariate analyzes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PAF and experience of symptomatic atrial fibrillation verified by ECG in the last six months

Exclusion Criteria:

* language difficulties, multi-diagnosis and/or cognitive dysfunction (eg, diagnoses of mental illness, dementia) who are judged not to be able to perform yoga. Individuals with persistent or permanent atrial fibrillation are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of paroxysmal atrial fibrillation will be identified from the list of patients scheduled for second visits at the Arrhythmia Polyclinic ("Arytmimottagningen") at the Cardiology Clinic, Danderyd Hospital. The selection will also be made from other hospitals in the Stockholm County Council.
Sampling Method: Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | Three months

SECONDARY OUTCOMES:
heart rate variability | three months

OTHER OUTCOMES:
Episodes of arrythmia is decreasing | three months

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rydell-Karlsson, RN, PhD, Principal Investigator — Sophiahemmet University, Stockholm
Locations (1):
- Karolinska Institute Danderyd hospital, Stockholm, Sweden